CLINICAL TRIAL: NCT02098343
Title: PiSARRO: p53 Suppressor Activation in Recurrent High Grade Serous Ovarian Cancer, a Phase Ib/II Study of Systemic Carboplatin Combination Chemotherapy With or Without APR-246
Brief Title: p53 Suppressor Activation in Recurrent High Grade Serous Ovarian Cancer, a Phase Ib/II Study of Systemic Carboplatin Combination Chemotherapy With or Without APR-246
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APR-407
Record Dates: First submitted 2014-03-19; First posted 2014-03-28 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Platinum Sensitive Recurrent High-grade Serous Ovarian Cancer With Mutated p53
Keywords: Ovarian cancer; Ovarian carcinoma; High Grade Serous Ovarian Cancer; Recurrent Cancer; Resistant Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — eprenetapopt; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Phase Ib. APR-246 (35mg/kg) + Carboplatin/PLD. (Experimental): Dose escalation of APR-246.
  Interventions: Drug: APR-246; Drug: Carboplatin and Pegylated Liposomal Doxorubicin Hydrochloride (PLD)
- Phase II: Arm A. APR-246 + Carboplatin/PLD. (Experimental): Experimental
  Interventions: Drug: APR-246; Drug: Carboplatin and Pegylated Liposomal Doxorubicin Hydrochloride (PLD)
- Phase II: Arm B. Carboplatin/PLD. (Active Comparator): Active Comparator
  Interventions: Drug: Carboplatin and Pegylated Liposomal Doxorubicin Hydrochloride (PLD)
- Phase Ib. APR-246 (50mg/kg) + Carboplatin/PLD. (Experimental): Dose escalation of APR-246.
  Interventions: Drug: APR-246; Drug: Carboplatin and Pegylated Liposomal Doxorubicin Hydrochloride (PLD)
- Phase Ib. APR-246 (67.5mg/kg) + Carboplatin/PLD. (Experimental): Dose escalation of APR-246.
  Interventions: Drug: APR-246; Drug: Carboplatin and Pegylated Liposomal Doxorubicin Hydrochloride (PLD)

INTERVENTIONS:
Drug: APR-246 — Intravenous infusion.
  Arms: Phase II: Arm A. APR-246 + Carboplatin/PLD.; Phase Ib. APR-246 (35mg/kg) + Carboplatin/PLD.; Phase Ib. APR-246 (50mg/kg) + Carboplatin/PLD.; Phase Ib. APR-246 (67.5mg/kg) + Carboplatin/PLD.
Drug: Carboplatin and Pegylated Liposomal Doxorubicin Hydrochloride (PLD) — Intravenous infusion.

SUMMARY:
The purpose of this study is to make a preliminary assessment of the efficacy of a combined APR-246 and carboplatin/PLD chemotherapy regimen, compared with carboplatin/PLD chemotherapy regimen alone, in patients with platinum sensitive recurrent high grade serous ovarian cancer (HGSOC) with mutated p53. In addition, the study aims to assess the safety profile of the combined APR-246 and carboplatin/PLD chemotherapy regimen compared with carboplatin/PLD chemotherapy regimen alone, to evaluate potential biomarkers, and to assess the biological activity in tumor and surrogate tissues. The trial will enroll up to a maximum of 400 patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed High Grade Serous Ovarian Cancer, and positive nuclear immunohistochemical (IHC) staining for p53
* Disease Progression between 6-24 months after a first or second platinum based regimen
* At least a single measurable lesion. Phase II patients only
* Adequate organ function prior to registration
* Toxicities from previous cancer therapies must have recovered to grade 1 (defined by Common Terminology Criteria for Adverse Events [CTCAE] 4.0) Chronic stable grade 2 peripheral neuropathy secondary to neurotoxicity from prior therapies may be considered on a case by case basis
* ECOG performance status of 0 to 1

Exclusion Criteria:

* Prior exposure to cumulative doses of doxorubicin >400 mg/m2 or epirubicin >720 mg/m2
* History of allergic reactions to carboplatin, platinum containing compounds or mannitol and/or hypersensitivity to PLD or to any of the excipients
* Unable to undergo imaging by either CT scan or MRI
* Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, neurological conditions, physical examination or laboratory findings) that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment related complications
* Concurrent malignancy requiring therapy (excluding non-invasive carcinoma or carcinoma in situ)
* Is taking concurrent (or within 4 week prior to registration) chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy that is considered to be investigational (i.e., used for non-approved indications(s) and in the context of a research investigation). Supportive care measures are allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (15):
  - UCLA, Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Oregon Health & Science University, Portland, Oregon
  - The University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Parkland, UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Massey Cancer Center, Virginia Commonwealth University, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
- Belgium (5):
  - Antwerp University Hospital, Antwerp
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - Medische oncologie, Universitair Ziekenhuis Gent, Ghent
  - Leuven University Hospitals, Leuven
- France (7):
  - Centre Léon Bérard, Lyon
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre Catherine de Sienne, Nantes
  - Institut Curie, Paris
  - Hôpital des Diaconesses (Site Reuilly), Paris
  - Centre Paul Strass, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Germany (5):
  - Praxisklinik, Krebsheilkunde für Frauen, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsfrauenklinik Ulm, Ulm
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
- Spain (11):
  - Institut Català d'Oncologia, Hospital Germans Trias i Pujol, Badalona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Centro Oncologico MD Anderson, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Araba, Vitoria-Gasteiz
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (7):
  - Bristol Haematology & Oncology Centre, University Hospitals Bristol, Bristol
  - Cambridge Cancer Trials Centre, Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital, Cambridge
  - Edinburgh Cancer Research Centre, The University of Edinburgh, Edinburgh
  - The Clatterbridge Cancer Center NHS Foundation Trust, Liverpool
  - The Royal Marsden NHS Foundation Trust, London
  - Imperial College London, Hammersmith Hospital Campus, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Background] Lehmann S, Bykov VJ, Ali D, Andren O, Cherif H, Tidefelt U, Uggla B, Yachnin J, Juliusson G, Moshfegh A, Paul C, Wiman KG, Andersson PO. Targeting p53 in vivo: a first-in-human study with p53-targeting compound APR-246 in refractory hematologic malignancies and prostate cancer. J Clin Oncol. 2012 Oct 10;30(29):3633-9. doi: 10.1200/JCO.2011.40.7783. Epub 2012 Sep 10. PMID 22965953
- [Background] Deneberg S, Cherif H, Lazarevic V, Andersson PO, von Euler M, Juliusson G, Lehmann S. An open-label phase I dose-finding study of APR-246 in hematological malignancies. Blood Cancer J. 2016 Jul 15;6(7):e447. doi: 10.1038/bcj.2016.60. No abstract available. PMID 27421096
- See also: Aprea Therapeutics AB's website (Sponsor) — http://www.aprea.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase Ib. APR-246 (35mg/kg) + Carboplatin/PLD. | Phase Ib. APR-246 (50mg/kg) + Carboplatin/PLD. | Phase Ib. APR-246 (67.5mg/kg) + Carboplatin/PLD. | Phase II: Arm A. APR-246 + Carboplatin/PLD. | Phase II: Arm B. Carboplatin/PLD.
Started | 9 | 6 | 21 | 105 | 106
Completed | 9 | 6 | 20 | 105 | 106
Not Completed | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 36 pts in Ph1b, and 211 patients in Ph2 were enrolled. One patient from the 67.5 mg/kg dose cohort was withdrawn from the study prior to initiating treatment. Another patient in the 67.5 mg/kg dose cohort did not meet the eligibility criteria (Exclusion criteria). The eligibility issue for this patient was discovered after the patient had commenced treatment. However, the patient continued the study treatment since it would have been unethical to withdraw the patient from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ib. APR-246 (35mg/kg) + Carboplatin/PLD. | Phase Ib. APR-246 (50mg/kg) + Carboplatin/PLD. | Phase Ib. APR-246 (67.5mg/kg) + Carboplatin/PLD. | Phase II: Arm A. APR-246 + Carboplatin/PLD. | Phase II: Arm B. Carboplatin/PLD. | Total
Number analyzed (Participants) | 9 | 6 | 20 | 105 | 106 | 246
Age, Categorical [Count of Participants; unit: Participants] — Population: 36 patients were enrolled in the Phase Ib study. One patient from the 67.5 mg/kg dose cohort was withdrawn from the study prior to initiating APR-246 treatment due to Investigator's decision.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 5 | 4 | 10 | 69 | 57 | 145
    >=65 years | 4 | 2 | 10 | 36 | 49 | 101
Age, Continuous [Median (Full Range); unit: years] | 63 [47 to 71] | 62 [48 to 75] | 64.5 [47 to 78] | 61 [31 to 80] | 64 [37 to 88] | 62 [31 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 20 | 105 | 106 | 246
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One patient in the 67.5 mg/kg dose cohort (Patient 441-P016) did not meet the eligibility criteria (Exclusion criteria). The eligibility issue for this patient was discovered after the patient had commenced treatment. However, the patient continued the study treatment since it would have been unethical to withdraw the patient from the study.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 3 | 3 | 2 | 8
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 1 | 1 | 2
    White | 9 | 6 | 17 | 88 | 81 | 201
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 13 | 22 | 35
Region of Enrollment [Number; unit: participants] — Population: One patient in the 67.5 mg/kg dose cohort (Patient 441-P016) did not meet the eligibility criteria (Exclusion criteria). The eligibility issue for this patient was discovered after the patient had commenced treatment. However, the patient continued the study treatment since it would have been unethical to withdraw the patient from the study.
  participants
    Netherlands | 0 | 0 | 0 | 12 | 2 | 14
    Sweden | 0 | 0 | 0 | 1 | 3 | 4
    Belgium | 2 | 1 | 4 | 10 | 10 | 27
    United States | 0 | 0 | 0 | 17 | 20 | 37
    United Kingdom | 7 | 5 | 16 | 33 | 19 | 80
    France | 0 | 0 | 0 | 12 | 20 | 32
    Germany | 0 | 0 | 0 | 1 | 10 | 11
    Spain | 0 | 0 | 0 | 19 | 22 | 41

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Dose-limiting Toxicities (DLT) (See Description) of Combined APR-246 and Carboplatin/PLD Regimen
Description: DLT: Hematological and non-hematological toxicities according to grade/days stated in the protocol.
Time Frame: Until the end of the first treatment cycle, i.e., Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib. APR-246 (35mg/kg) + Carboplatin/PLD. | Phase Ib. APR-246 (50mg/kg) + Carboplatin/PLD. | Phase Ib. APR-246 (67.5mg/kg) + Carboplatin/PLD.
Number analyzed (Participants) | 9 | 6 | 20
Participants | 0 | 1 | 0

2. Primary Outcome: Phase Ib and II: Progression Free Survival (PFS)
Description: Phase Ib: Progression-free Survival is calculated from date of enrollment to the date of disease progression or death due to any cause, whichever occurs first. Symptomatic deterioration is not considered PD. For a patient without evidence of disease progression or death, Progression-free survival will be censored at the date of last evaluable tumor assessment. Patients with no evaluable tumor assessments will be censored at the date of first study drug administration.
  Phase II: Progression-free survival (PFS) based on Blinded Independent Central Review (BICR) is the primary endpoint and is defined as the number of days from the date of randomization to the date of objective disease progression or relapse (according to RECIST v1.1 only) or death due to any cause, whichever occurs first. If neither event occurs, PFS is censored at the date of the last evaluable tumor assessment. Symptomatic deterioration is not considered objective disease progression.
Time Frame: Up to 24 months
Population: Ph Ib = Efficacy Evaluable
  Ph II = ITT
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase Ib. APR-246 (35mg/kg) + Carboplatin/PLD. | Phase Ib. APR-246 (50mg/kg) + Carboplatin/PLD. | Phase Ib. APR-246 (67.5mg/kg) + Carboplatin/PLD. | Phase II: Arm A. APR-246 + Carboplatin/PLD. | Phase II: Arm B. Carboplatin/PLD.
Number analyzed (Participants) | 7 | 4 | 19 | 105 | 106
days | 330 [280 to 444] | 277.5 [175 to 375] | 313 [98 to 590] | 283 [240 to 314] | 295 [259 to 335]

3. Secondary Outcome: Phase Ib and Phase II: Overall Response Rate (RR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 24 months
Population: Phase Ib = Efficacy Evaluable population
  Phase II = ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Phase Ib. APR-246 + Carboplatin/PLD.; Phase Ib. APR-246 (50mg/kg) + Carboplatin/PLD.; Phase Ib. APR-246 (67.5mg/kg) + Carboplatin/PLD.: Dose escalation of APR-246.
  APR-246: Intravenous infusion.
  Carboplatin and Pegylated Liposomal Doxorubicin Hydrochloride (PLD): Intravenous infusion.
Arm/Group | Phase Ib. APR-246 + Carboplatin/PLD. | Phase Ib. APR-246 (50mg/kg) + Carboplatin/PLD. | Phase Ib. APR-246 (67.5mg/kg) + Carboplatin/PLD. | Phase II: Arm A. APR-246 + Carboplatin/PLD. | Phase II: Arm B. Carboplatin/PLD.
Number analyzed (Participants) | 7 | 4 | 19 | 105 | 106
Participants
  Complete Response (CR) | 1 | 0 | 2 | 10 | 3
  Partial response (PR) | 5 | 1 | 9 | 42 | 50
  Stable Disease (SD) | 1 | 3 | 5 | 27 | 37
  Progressive Disease (PD) | 0 | 0 | 0 | 15 | 5
  Not Evaluable (NE) | 0 | 0 | 3 | 11 | 11

ADVERSE EVENTS:
Time Frame: TEAEs were defined as events occurring on or after Day 1 Cycle 1 up to and including 30 days after last dose, or Cycle 6, up to 7 months.
Description: Ph1b: All dose groups in Ph1b are combined and reported together due to small numbers in escalation phase:
  n=9 at 35mg/kg n=6 at 50mg/kg n=20 at 67.5mg/kg
  Ph2: Safety evaluable population is defined as all randomized patients who received any amount of study medication [APR-246, carboplatin, or PLD], regardless of duration of treatment.
Groups:
- Phase Ib. APR-246 (35mg/kg) + Carboplatin/PLD.; Phase Ib. APR-246 (50mg/kg) + Carboplatin/PLD.; Phase Ib. APR-246 (67.5mg/kg) + Carboplatin/PLD.: Dose escalation of APR-246.
  APR-246: Intravenous infusion.
  Carboplatin and Pegylated Liposomal Doxorubicin Hydrochloride (PLD): Intravenous infusion.
  All dose groups in Ph1b are combined and reported together due to small numbers in escalation phase:
  n=9 at 35mg/kg n=6 at 50mg/kg n=20 at 67.5mg/kg
Arm/Group | Phase Ib. APR-246 (35mg/kg) + Carboplatin/PLD. | Phase Ib. APR-246 (50mg/kg) + Carboplatin/PLD. | Phase Ib. APR-246 (67.5mg/kg) + Carboplatin/PLD. | Phase II: Arm A. APR-246 + Carboplatin/PLD. | Phase II: Arm B. Carboplatin/PLD.
All-Cause Mortality (participants affected / at risk) | 4/9 | 3/6 | 10/20 | 0/99 | 2/101
Serious Adverse Events (participants affected / at risk) | 3/9 | 4/6 | 12/20 | 31/99 | 17/101
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6 | 20/20 | 99/99 | 101/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib. APR-246 (35mg/kg) + Carboplatin/PLD. (N=9) | Phase Ib. APR-246 (50mg/kg) + Carboplatin/PLD. (N=6) | Phase Ib. APR-246 (67.5mg/kg) + Carboplatin/PLD. (N=20) | Phase II: Arm A. APR-246 + Carboplatin/PLD. (N=99) | Phase II: Arm B. Carboplatin/PLD. (N=101)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 4 | 4
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Vomitting (Gastrointestinal disorders) | 0 | 0 | 6 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 2 | 3 | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Phlebitis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib. APR-246 (35mg/kg) + Carboplatin/PLD. (N=9) | Phase Ib. APR-246 (50mg/kg) + Carboplatin/PLD. (N=6) | Phase Ib. APR-246 (67.5mg/kg) + Carboplatin/PLD. (N=20) | Phase II: Arm A. APR-246 + Carboplatin/PLD. (N=99) | Phase II: Arm B. Carboplatin/PLD. (N=101)
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 4 | 12 | 11
Nausea (Gastrointestinal disorders) | 8 | 3 | 16 | 67 | 57
Vomitting (Gastrointestinal disorders) | 4 | 2 | 16 | 42 | 23
Diarrhea (Gastrointestinal disorders) | 3 | 4 | 10 | 12 | 16
Constipation (Gastrointestinal disorders) | 5 | 3 | 8 | 36 | 33
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 6 | 16 | 16
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 3 | 8 | 6
Asthenia (General disorders) | 0 | 0 | 0 | 19 | 22
Fatigue (General disorders) | 8 | 5 | 16 | 47 | 38
Mucosal inflammation (General disorders) | 4 | 1 | 5 | 20 | 22
Pyrexia (General disorders) | 0 | 1 | 6 | 13 | 10
Device occlusion (General disorders) | 2 | 2 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 6 | 3 | 15 | 42 | 5
Headache (Nervous system disorders) | 7 | 3 | 6 | 16 | 11
Dysgeusia (Nervous system disorders) | 6 | 3 | 3 | 3 | 6
Tremor (Nervous system disorders) | 1 | 1 | 3 | 8 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 4 | 11 | 6
Neutropenia (Blood and lymphatic system disorders) | 7 | 6 | 15 | 56 | 39
Anemia (Blood and lymphatic system disorders) | 3 | 3 | 6 | 31 | 30
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 6 | 23 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5 | 13 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 10 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2 | 2
Device related infection (Infections and infestations) | 1 | 2 | 3 | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 0 | 4 | 10 | 18
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 9 | 19 | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 12 | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 11 | 18
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 4 | 10 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 6 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 15 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 16 | 4
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 12 | 11
Platelet count decreased (Investigations) | 0 | 0 | 0 | 11 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 3 | 5 | 6
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 4 | 4
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 5 | 5
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 7 | 1
Chills (General disorders) | 0 | 0 | 3 | 3 | 2
Infusion site erythema (General disorders) | 0 | 0 | 2 | 2 | 1
Oedema peripheral (General disorders) | 0 | 0 | 2 | 7 | 3
Malaise (General disorders) | 0 | 0 | 1 | 5 | 2
Dyskinesia (Nervous system disorders) | 0 | 0 | 3 | 3 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 2 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 2 | 3 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 8 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 6 | 3
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 8 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 5 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 5 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 6 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 3 | 2 | 1
Infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Infusion site infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 2 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 5 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 6 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 5 | 7
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 7
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 2 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 3 | 2 | 10
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 4 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 2 | 3 | 3
Weight decreased (Investigations) | 0 | 0 | 3 | 2 | 3
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 7 | 5
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2 | 4
Flushing (Vascular disorders) | 0 | 0 | 2 | 5 | 2
Palpitations (Vascular disorders) | 0 | 0 | 3 | 4 | 0
Photophobia (Eye disorders) | 0 | 0 | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2 | 2 | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 9 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 7 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT02098343/Prot_SAP_000.pdf